CLINICAL TRIAL: NCT02084901
Title: Comparison of Biodegradable Stents: Orsiro and BioMatrix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2013-0083
Record Dates: First submitted 2014-03-09; First posted 2014-03-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: All-comer; Percutaneous Coronary Intervention
Keywords: Biodegradable stents; converage; OCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orsiro Arm (Experimental)
  Interventions: Device: Drug-eluting biodegradable stent Orsiro implantation
- BioMatrix or BioMatrix Flex Arm (Active Comparator)
  Interventions: Device: Drug-eluting biodegradable stent BioMatrix or BioMatrix Flex implantation

INTERVENTIONS:
Device: Drug-eluting biodegradable stent Orsiro implantation — Drug-eluting biodegradable stent Orsiro implantation
  Arms: Orsiro Arm
Device: Drug-eluting biodegradable stent BioMatrix or BioMatrix Flex implantation — Drug-eluting biodegradable stent BioMatrix or BioMatrix Flex implantation
  Arms: BioMatrix or BioMatrix Flex Arm

SUMMARY:
The use of a biodegradable polymer has the potential to reduce the sustained inflammatory response of the arterial wall, facilitating re-endothelialization and minimizing the risk of thrombus formation and late restenosis. In the study, we are going to two biodegradable polymer stents, Orsiro and BioMatrix, especially regarding the stent strut coverage by optical coherence tomography at 3 months after stent implantation.

The primary objective of this study is to test the hypothesis that Orsiro is non-inferior to Biomatrix in terms of stent strut coverage by optical coherence tomography at 3 months. The secondary endpoint is clinical outcomes up to 1 year.

DETAILED DESCRIPTION:
The use of a biodegradable polymer has the potential to reduce the sustained inflammatory response of the arterial wall, facilitating re-endothelialization and minimizing the risk of thrombus formation and late restenosis. In the study, we are going to two biodegradable polymer stents, Orsiro and BioMatrix, especially regarding the stent strut coverage by optical coherence tomography at 3 months after stent implantation.

The primary objective of this study is to test the hypothesis that Orsiro is non-inferior to Biomatrix in terms of stent strut coverage by optical coherence tomography at 3 months. The secondary endpoint is clinical outcomes up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 20 years old
2. Patients in the treatment of subjects with all-comer who are to undergo PCI

Exclusion Criteria:

1. Pregnant women or women with potential childbearing
2. Life expectancy < 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Neointimal coverage at 3 month after stent implantation | At 3 months after stent implantation
  The percentage of stent uncoverage measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seodaemun-gu, Shinchondong, Seoul, South Korea